CLINICAL TRIAL: NCT06067607
Title: Examining the Effect of Eye Gaze Technology on Children With Cortical Visual Impairment and Its Impact on Occupational Performance
Brief Title: Examining the Effect of Eye Gaze Technology on Children With Cortical Visual Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rockhurst University (Other)
Responsible Party: Principal Investigator, Tammy Bruegger, Assistant Professor of Occupational Therapy, Rockhurst University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-09
Record Dates: First submitted 2023-03-27; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Cortical/Cerebral Visual Impairment; Cerebral Palsy
Keywords: Cortical/Cerebral Visual Impairment; Vision; Occupational Performance; Sensory Processing
MeSH Terms: conditions — Blindness, Cortical; Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Mixed Design, Pre/Post Pre-Experimental Design
Masking Description: Masking is not used as this is not a randomized control study and because eye gaze software will objectively document improvements in visual abilities. Scoring on COPM will be conducted by separate investigator from the CVI Range.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eye gaze technology intervention (Experimental): Participants will use eye gaze technology and software activities as an intervention to improve visual abilities.
  Interventions: Other: eye gaze technology

INTERVENTIONS:
Other: eye gaze technology — eye gaze technology and software activities

SUMMARY:
The goal of this study is to learn about eye gaze technology's use as an assessment and intervention of visual skills and the impact on occupational performance in children with cortical/cerebral visual impairment. The main questions the study aims to answer are:

* Does the use of eye gaze technology with graded visual activities improve visual abilities:
* Does an improvement in visual abilities improve occupational performance? - What are the factors that correlate with improved visual abilities?

Participants will complete the Pre-test with Canadian Occupational Performance Measurement, Cortical Visual Impairment Range, Sensory Profile and Sensory Processing Checklist for Children with Visual Impairment. Then will participate in eye gaze technology activities using eye gaze software with graded visual games for 20 minutes per day for 4 weeks. Observations of positioning, head/eye position, sensory processing, and types of eye gaze activities used during the session. Pre test, daily and post test percentage scores on the eye gaze activities will be recorded. Then the child will complete post testing with the Canadian Occupational Performance Measurement and Cortical Visual Impairment Range.

DETAILED DESCRIPTION:
Approval to perform this study was granted by the Rockhurst University Institutional Review Board (IRB) and the Rockhurst University (RU) Occupational Therapy Department prior to participant recruitment. Written informed consent was obtained from the parents of the participants and physical assent was obtained from the children older than 8 years of age. Researchers were trained by the primary investigator following an established written protocol for eye gaze technology administration. The protocal involved set up of the eye gaze camera and laptop computer with calibration of the camera to the child's eyes using Gaze Point software by Tobii. If the camera is unable to be calibrated to the child's eyes it will be calibrated with the therapists eyes in the same position as the child with eyes centered in the middle of the calibration screen. The child will be positioned 15-18 inches from the screen with a black trifold board behind the screen and lights turned off in a quiet room to decrease distractions. Teachers and therapists involved with data collection were trained in eye gaze technology administration following the protocal. Data was collected by the Insight and Learning Curve eye gaze software using percentage scoring and a heat map/line plot pictures. Eye gaze technology sessions will last 20 minutes, three to five days per week, for four weeks. Images presented during the eye gaze sessions include the following characteristics: single colors, reduced complexity, movement of the image, reduced surrounding auditory and visual clutter, and reduced inclusion of multiple colors. Demographic information, Canadian Occupational Performance Measurement (COPM,) Cortical Visual Impairment (CVI) Range, Sensory Profile Short Form (SP), and Sensory Processing Checklist for Children with Visual Impairment (SPCCVI) scores were collected by the researchers prior to administration of the eye gaze intervention. A baseline score was obtained from the Insight software using a mean of the subtests completed and then a mean of the subtests 4 weeks later. Scores for all of the measures except for the Sensory Profile and SPCCVI were then re-collected 4 weeks later at the conclusion of the study. Data was compiled and stored on a file on a password protected computer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Cortical/Cerebral Visual Impairment by Physician
* 2-10 years of age
* Parent or Caregiver available for interview

Exclusion Criteria:

* Only ocular visual impairment,
* Age above 10 years of age.
* No parent or caregiver available for interview

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-04-05 (Estimated); Study Completion 2024-04-05 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measurement (COPM) | Measure change from baseline and after 4 weeks of intervention.
  semi structured interview of daily function and occupational performance using score for importance, performance and satisfaction of occupational performance skills. Minimum score of 0-10, 10 being maximum score. Increased score shows higher performance, and satisfaction.
Eye Gaze Technology Software Scoring: Insight Software | Measure change from baseline and after 4 weeks of intervention.
  Computerized score of visual abilities conducted by software and eye gaze camera. Scale of 0-100%. Increased percentage score shows improvement in eye gaze skill.
Cortical Visual Impairment Range (CVI) | Measure change from baseline and after 4 weeks of intervention.
  Test of functional vision and visual processing. Scale of 0-10 on CVI Range scores range from 0 to 10, with 10 indicating the best functional vision. The scores are further divided into three phases (phase I: 0-3, phase II: 4-7 and phase III: 8-10. Severity of each visual behavior is rated on 0-1 scale. 1 means that behavior has resolved and is no longer observed.

OTHER OUTCOMES:
Sensory Processing Checklist for Children with Visual Impairment (SPCCVI) | Test given at baseline.
  Caregiver checklist of observed behaviors of sensory processing.SPCCVI scores on 0-5 scale with 0 indicating sensory behavior not seen and 5 indicating behavior "always observed". Higher scores relate to increased sensory processing behaviors.
Sensory Profile-Short Form (SPSF) | Test given at baseline.
  Caregiver Test of sensory processing. The rating scale on the Sensory Profile ranges from 1 (Almost Never) to 5 (Almost Always), with higher scores indicating a higher frequency of specific sensory responses.

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Bruegger, Principal Investigator — Rockhurst University
Locations (1):
- The Children's Center for the Visually Impaired, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fazzi E, Micheletti S, Calza S, Merabet L, Rossi A, Galli J; Early Visual Intervention Study Group. Early visual training and environmental adaptation for infants with visual impairment. Dev Med Child Neurol. 2021 Oct;63(10):1180-1193. doi: 10.1111/dmcn.14865. Epub 2021 May 4. PMID 34813110
- [Background] Rowe FJ, Hanna K, Evans JR, Noonan CP, Garcia-Finana M, Dodridge CS, Howard C, Jarvis KA, MacDiarmid SL, Maan T, North L, Rodgers H. Interventions for eye movement disorders due to acquired brain injury. Cochrane Database Syst Rev. 2018 Mar 5;3(3):CD011290. doi: 10.1002/14651858.CD011290.pub2. PMID 29505103
- [Background] Lammers NA, Van den Berg NS, Lugtmeijer S, Smits AR, Pinto Y, de Haan EHF; visual brain group. Mid-range visual deficits after stroke: Prevalence and co-occurrence. PLoS One. 2022 Apr 1;17(4):e0262886. doi: 10.1371/journal.pone.0262886. eCollection 2022. PMID 35363793
- [Background] Vancleef K, Janssens E, Petre Y, Wagemans J, Ortibus E. Assessment tool for visual perception deficits in cerebral visual impairment: development and normative data of typically developing children. Dev Med Child Neurol. 2020 Jan;62(1):111-117. doi: 10.1111/dmcn.14303. Epub 2019 Jul 2. PMID 31267521
- [Background] Bennett, C. R., Bailin, E. S., Gottlieb, T. K., Bauer, C. M., Bex, P. J., & Merabet, L. B. (2018). Virtual reality based assessment of static object visual search in ocular compared to cerebral visual impairment. In International Conference on Universal Access in Human-Computer Interaction (pp. 28-38). Springer, Cham. https://doi.org/10.1007/978-3-319-92052-8_3
- [Background] Manley CE, Bennett CR, Merabet LB. Assessing Higher-Order Visual Processing in Cerebral Visual Impairment Using Naturalistic Virtual-Reality-Based Visual Search Tasks. Children (Basel). 2022 Jul 26;9(8):1114. doi: 10.3390/children9081114. PMID 35892617
- [Background] Ben Itzhak N, Kooiker MJG, van der Steen J, Pel JJM, Wagemans J, Ortibus E. The relation between visual orienting functions, daily visual behaviour and visuoperceptual performance in children with (suspected) cerebral visual impairment. Res Dev Disabil. 2021 Dec;119:104092. doi: 10.1016/j.ridd.2021.104092. Epub 2021 Oct 5. PMID 34619456
- [Background] Ferziger, N. (2017). Assessment of gaze responses of children with Cerebral Palsy and cerebral visual impairment: Implementation of a computerized video coding system. The American Journal of Occupational Therapy, 71(4_Supplement_1). https://doi.org/10.5014/ajot.2017.71s1-po1138
- [Background] VerMaas-Hannan, J., Gehringer, J., Wilson, T., & Kurz, M. (2019). Visual motion perception is aberrant in children with cerebral palsy. The American Journal of Occupational Therapy, 73(4_Supplement_1). https://doi.org/10.5014/ajot.2019.73s1-rp302b
- [Background] Cemali M, Pekcetin S, Aki E. The Effectiveness of Sensory Integration Interventions on Motor and Sensory Functions in Infants with Cortical Vision Impairment and Cerebral Palsy: A Single Blind Randomized Controlled Trial. Children (Basel). 2022 Jul 27;9(8):1123. doi: 10.3390/children9081123. PMID 36010014
- [Background] Galli J, Loi E, Molinaro A, Calza S, Franzoni A, Micheletti S, Rossi A, Semeraro F, Fazzi E; CP Collaborative Group. Age-Related Effects on the Spectrum of Cerebral Visual Impairment in Children With Cerebral Palsy. Front Hum Neurosci. 2022 Mar 2;16:750464. doi: 10.3389/fnhum.2022.750464. eCollection 2022. PMID 35308614
- [Background] Kovarski K, Caetta F, Mermillod M, Peyrin C, Perez C, Granjon L, Delorme R, Cartigny A, Zalla T, Chokron S. Emotional face recognition in autism and in cerebral visual impairments: In search for specificity. J Neuropsychol. 2021 Jun;15(2):235-252. doi: 10.1111/jnp.12221. Epub 2020 Sep 13. PMID 32920927
- [Background] Racey C, Franklin A, Bird CM. The processing of color preference in the brain. Neuroimage. 2019 May 1;191:529-536. doi: 10.1016/j.neuroimage.2019.02.041. Epub 2019 Feb 21. PMID 30798014
- [Background] Chang MY, Borchert MS. Methods of visual assessment in children with cortical visual impairment. Curr Opin Neurol. 2021 Feb 1;34(1):89-96. doi: 10.1097/WCO.0000000000000877. PMID 33230032
- [Background] Chang MY, Borchert MS. Advances in the evaluation and management of cortical/cerebral visual impairment in children. Surv Ophthalmol. 2020 Nov-Dec;65(6):708-724. doi: 10.1016/j.survophthal.2020.03.001. Epub 2020 Mar 19. PMID 32199940
- [Background] Kran BS, Lawrence L, Mayer DL, Heidary G. Cerebral/Cortical Visual Impairment: A Need to Reassess Current Definitions of Visual Impairment and Blindness. Semin Pediatr Neurol. 2019 Oct;31:25-29. doi: 10.1016/j.spen.2019.05.005. Epub 2019 May 11. PMID 31548020
- [Background] Gartz, R., Dickerson, A., & Radloff, J. (2019). Effectiveness of visual scanning compensatory training after stroke. The American Journal of Occupational Therapy, 73(4_Supplement_1). https://doi.org/10.5014/ajot.2019.73s1-po2039